CLINICAL TRIAL: NCT02862977
Title: Phase III, National, Multicenter, Randomized, Double-blind, Double-masked, Compare the Efficacy of Ketoprofen, Cyclobenzaprine and Caffeine Association Versus Cyclobenzaprine and Caffeine (Miosan Caf®) in the Treatment of Osteomuscular Pain in Adults
Brief Title: Efficacy and Safety of the Combination of Ketoprofen and Cyclobenzaprine and Caffeine in Osteomuscular Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS1415
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Ketoprofen; Caffeine; cyclobenzaprine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMS association (Experimental): The patient will take 2 tablets (combination of ketoprofen and cyclobenzaprine and caffeine), oral, per day, each 12h.
  Interventions: Drug: ketoprofen and cyclobenzaprine association with caffeine
- Miosan Caf® (Active Comparator): The patient will take 2 tablets (combination of Cyclobenzaprine and caffeine), oral, per day, each 12h.
  Interventions: Drug: Cyclobenzaprine with caffeine

INTERVENTIONS:
Drug: ketoprofen and cyclobenzaprine association with caffeine — The patient will take 2 tablets (combination of ketoprofen and cyclobenzaprine and caffeine), oral, per day, each 12h
  Other Names: EMS association
  Arms: EMS association
Drug: Cyclobenzaprine with caffeine — The patient will take 2 tablets (combination of cyclobenzaprine and caffeine), oral, per day, each 12h
  Other Names: Miosan Caf®
  Arms: Miosan Caf®

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of an association with one anti-inflammatory and one muscle relaxant plus caffeine compared to one anti-inflammatory plus caffeine in the treatment of osteomuscular pain in adults.

DETAILED DESCRIPTION:
* Double-blind,randomized, multicenter
* Maximal experiment duration: 9 days
* 02 or 03 visits and a phone contact
* Evaluate the efficacy of an association with one anti-inflammatory and one muscle relaxant agent with caffeine compared to the one muscle relaxant agent plus caffeine in the treatment of osteomuscular pain in adults.
* Adverse events evaluation

ELIGIBILITY:
Inclusion Criteria:

* Signed Consent of the patient;
* Participants presenting musculoskeletal pain, moderate or moderately severe, with VAS (visual analog scale) greater than 40 mm for a period of less than seven (7) days.

Exclusion Criteria:

* Patients with any clinically significant disease that in the investigator is opinion can´t participate in the study;
* Patients with any laboratory finding or image finding that in the investigator is opinion can´t participate in the clinical trial;
* Patients with history of hypersensitivity to any of the formula compounds;
* Participation in clinical trial in the year prior to this study;
* Pregnancy or risk of pregnancy and lactating patients;
* Patients who were in use of drugs that can interfere with evaluation;
* History of with rheumatic diseases, fibromyalgia, osteoarticular diseases, dystonia, dystrophies and myopathies, acute infectious diseases, gastric duodenal ulcer or gastritis;
* Renal or hepatic impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of osteomuscular treatment based on proportion of participants who achieve the 2, 3 or 4 points in the pain scale. | 48 hours

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | Maximal experiment duration: 9 days

CONTACTS AND LOCATIONS:
Locations (6):
- Brazil (6):
  - Associação dos funcionários públicos do estado do RGS, Porto Alegre, Rio Grande do Sul
  - Centro de Medicina Reprodutiva Dr Carlos Isaia Filho, Porto Alegre, Rio Grande do Sul
  - Allegisa, Campinas, São Paulo
  - CECIP JAU - Centro De Estudos Clinicos do Interior Paulista, Jaú, São Paulo
  - Marcio Antonio Pereira Clinica de Endocrinologia, São José dos Campos, São Paulo
  - AFIP -Associação Fundo de Incentivo a Pesquisa, São Paulo, São Paulo